CLINICAL TRIAL: NCT06220045
Title: Comparison Between the Use of a Polypropylene (PP) Prophylactic Mesh and a Polyvinylidene Fluoride (PVDF) Mesh in the Closure of Midline Laparotomy in Emergency Colorectal Surgery for High-risk Patients of Incisional Hernia. Impact on Surgical Wound Infection.
Brief Title: Comparing PP and PVDF Meshes in Midline Laparotomy Closure for High-risk Colorectal Surgery. Impact on Incisional Hernia and Surgical Wound Infection.
Acronym: PROFIMESH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Responsible Party: Principal Investigator, Fernandez Zamora, Principal Investigator, Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023.226
Record Dates: First submitted 2024-01-11; First posted 2024-01-23 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Cancer; Wound Infection; Hernia Incisional
Keywords: Colorectal cancer; Wound Infection; Hernia Incisional; Mesh; Polypropylene; PVDF
MeSH Terms: conditions — Colorectal Neoplasms; Wound Infection; Incisional Hernia

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients meeting the inclusion criteria for the study will be randomized 1:1 using random number generation functions with SPSS v.21 software into either the PP or PVDF group. This randomization will be carried out using sealed opaque envelopes at the time immediately preceding the onset of the surgical intervention within the operating room. The envelope will be opened within the operating room once the closure of the midline laparotomy is initiated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polyvinylidene fluoride mesh (Experimental): In all patients, surgery will be performed according to their individual pathology. Once midline laparotomy closure is initiated, randomization will be conducted, and patients will be assigned to one of the two groups.
  PVDF Group (Polyvinylidene Fluoride Mesh): Midline laparotomy closure using the "small bites" technique associated with a prophylactic suprafascial polyvinylidene fluoride mesh
  Interventions: Combination Product: Polyvinylidene fluoride mesh
- Prophylactic polypropylene mesh (Experimental): In all patients, surgery will be performed according to their individual pathology. Once midline laparotomy closure is initiated, randomization will be conducted, and patients will be assigned to one of the two groups.
  PP Group (Polypropylene Mesh): Midline laparotomy closure using the "small bites" technique associated with a prophylactic suprafascial polypropylene mesh.
  Interventions: Combination Product: Prophylactic polypropylene mesh

INTERVENTIONS:
Combination Product: Polyvinylidene fluoride mesh — Midline laparotomy closure using the "small bites" technique associated with a prophylactic suprafascial polyvinylidene fluoride mesh.
  Arms: Polyvinylidene fluoride mesh
Combination Product: Prophylactic polypropylene mesh — Midline laparotomy closure using the "small bites" technique associated with a prophylactic suprafascial polypropylene mesh.
  Arms: Prophylactic polypropylene mesh

SUMMARY:
In the latest guidelines for abdominal wall closure in emergency surgery published in the World Journal of Emergency Surgery (WJES) in 2023, no specific recommendations are made in this regard.

Current literature does not provide any articles comparing these two types of mesh materials (PP vs PVDF) in emergency colorectal surgery. It is necessary to conduct a study comparing these two types of mesh materials, specifically in high-risk patients for incisional hernia and emergency colorectal surgery. This study aims to contribute to generating evidence regarding differences in wound infection incidence and potential subsequent complications, such as chronic pain.

It is essential to conduct a study comparing different methods of laparotomy closure, specifically in emergency colorectal surgery, to contribute valuable evidence regarding the incidence of incisional hernia and potential subsequent complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with colorectal pathology requiring urgent surgical treatment via midline laparotomy.
* Patients undergoing urgent laparoscopic surgery but requiring conversion to midline laparotomy.
* Need for urgent surgical treatment involving the colon and/or rectum, even in the presence of other abdominal pathologies.
* Age over 18 years.
* Signed informed consent (IC) from both the patient and the investigator
* Severe chronic obstructive pulmonary disease (COPD) according to the GOLD classification or decompensated COPD.
* BMI ≥ 35 kg/m2.
* Re-laparotomies.

Exclusion Criteria:

* Patients with psychiatric illnesses, addictions, or any disorder hindering the understanding of the Informed Consent.
* Inability to read or comprehend any of the languages in the Informed Consent (Catalan, Spanish).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of surgical wound infection | 30 postoperative days
  Compare the incidence of surgical wound infection between the two groups: Closure of midline laparotomy using the "small bites" technique associated with a suprafascial polypropylene mesh versus closure of midline laparotomy using the "small bites" technique associated with a suprafascial polyvinylidene fluoride mesh.

SECONDARY OUTCOMES:
Rate of incisional hernia | One year surgery
  Compare the rate of incisional hernia at one year post-surgery, postoperative complications, and abdominal pain at 6 and 12 months in both groups. Also, compare the rates of parastomal hernias.
Morbidity and mortality rates | 90 postoperative days
  Comparison between the two groups on various aspects related to postoperative morbidity and mortality. Other aspects to be evaluated include the time of initiation of tolerance to solid oral diet, onset of ambulation, presence of anastomotic dehiscence, need for reinterventions, and occurrence of complications according to the Clavien-Dindo classification at 30 and 90 days, as well as the mortality rate at 90 days. Additionally, the aim is to compare the rate of initiation of adjuvant treatment within the first 6 weeks post-surgery, if indicated.

CONTACTS AND LOCATIONS:
Locations (1):
- Colorectal Surgery Section, Department of General and Digestive Surgery, University Hospital of Girona,, Girona, Spain

IPD SHARING:
Plan to Share IPD: No